CLINICAL TRIAL: NCT04893603
Title: A Prospective, Multi-center, Single-arm Clinical Trial to Evaluate the Safety and Effectiveness of Transcatheter Aortic Valve System in Patients With Severe Aortic Stenosis With or Without Moderate or Lower Degree Regurgitation
Brief Title: To Evaluate Safety and Effectiveness of Transcatheter Aortic Valve System in Patients With Severe Aortic Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu Silara Meditech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Silara201901
Record Dates: First submitted 2021-04-28; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severe Aortic Valve Stenosis (Experimental): Patients will be treated with Transcatheter Aortic Valve Systerm
  Interventions: Device: Transcatheter Aortic Valve System

INTERVENTIONS:
Device: Transcatheter Aortic Valve System — Procedure: Transcatheter aortic valve replacement

SUMMARY:
To Evaluate the Safety and Effectiveness of Transcatheter Aortic Valve System ( Chengdu Silara Medtech Inc. ,Chengdu, China)in Patients with Severe Aortic Stenosis with or without Moderate or Lower Degree Regurgitation

DETAILED DESCRIPTION:
Transcatheter Aortic Valve System (Chengdu Silara Medtech Inc. ,Chengdu, China) will be used for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥70 years old;
2. Symptomatic severe aortic stenosis determined by echocardiogram, defined as: mean gradient ≥40 mmHg or peak jet velocity ≥4.0 m/s, or an aortic valve area <0.8 cm2 or aortic valve area index <0.5 cm2/m2.
3. NYHA Functional Class ≥II;
4. Life expectancy after aortic valve implantation thought to be >1 year;
5. Native valvular or peripheral vascular anatomy is appropriate for TAVR;
6. Patient is assessed by at least two cardiothoracic surgeons and recorded as not suitable for surgery;
7. Patient can understand the purpose of the study, voluntarily participates and signs the informed consent form and is willing to accept the relevant examination and clinical follow-up visits.

Exclusion Criteria:

1. Anatomy is not appropriate for percutaneous valve implantation. Native valve annulus diameter is not in the scope of application(native TAV diameter ≤21mm, or ≥30mm);
2. Evidence of an acute myocardial infarction within 30 days prior to the study procedure, defined as: Q-wave myocardial infarction, or non-Q-wave myocardial infarction, with CK-MB≥2 ULN/or elevated TN (WHO definition);
3. Any treatment for traumatic cardiac surgery within 30 day prior to the study procedure(except coronary revascularization);
4. Pre-existing prosthetic valve in any position(except severely dysfunctional aortic bioprosthesis), or severe (>3+) mitral insufficiency, or Gorlin syndrome;
5. Hematological abnormality, defined as: Leukopenia (WBC <3x10^9/L), acute anemia (Hb <90g/L), or thrombocytopenia (platelet count<50×109/L),history of bleeding diathesis or coagulopathy;
6. Hemodynamic unstable requiring myocardial contractile support or mechanical cardiac assistance;
7. Severe ventricular insufficiency. Left ventricular ejection fraction (LVEF) <20%;
8. Echocardiographic evidence of intra-cardiac thrombus or vegetation etc.;
9. Active pepticulcer or upper GI bleeding within 3 months prior to the study procedure;
10. Cerebral Vascular Accident (CVA) within 3 months prior to the study procedure, including TIA;
11. A known hypersensitivity or contraindication to aspirin, heparin, ticlopidine or clopidogrel, or sensitivity to contrast media, which cannot be adequately pre-medicated;
12. Patients with infective endocarditis or other active stage of infection;
13. Currently participating in an investigational drug or another device trial.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of All-cause Mortality | 12 months
  Percentage of subjects who died from all causes in this population.

SECONDARY OUTCOMES:
Rate of Device Success | Immediate post- procedure
  Device Success is defined as a composite of :
  1. Absence of procedural mortality AND
  2. Successful vascular access, delivery and deployment of the device, and successful retrieval of the delivery system AND
  3. Correct positioning of prosthetic heart valve into the proper anatomical location AND
  4. Intended performance of the prosthetic heart valve (mean aortic valve gradient<20 mmHg or peak velocity<3 m/s, and no severe prosthetic valve regurgitation or PVL)
Rate of Procedure Success | Immediate post- procedure
  Procedure Success is defined as no death, stroke, myocardial infarction and renal failure occurred within 72 hours after the operation on the basis of the final device success.
Delivery System Performance | Immediate post- procedure
  Delivery System Performance wil be evaluated subjectively by the researchers participating in the operation, which is generally classified as excellent, good ,average and poor.
Retrieval System Performance(if using) | Immediate post- procedure
  Retrieval System Performance wil be evaluated subjectively by the researchers participating in the operation, which is generally classified as excellent, good ,average and poor.
Exchange Systerm Evaluation | Immediate post- procedure
  Exchange Systerm Evaluation wil be evaluated subjectively by the researchers participating in the operation, which is generally classified as excellent, good ,average and poor.
Valvular function evaluation, including valve stenosis, AR, valve function(e.g. EOA, gradient) and PVL | Immediate post-procedure, 7days or discharge, 30 days, 6 months ,12months and 2-5 years
  The evaluation criteria refer to the 2012 edition of the Association for Valvular Academic Research (VARC-2) consensus document
Quality of Life Assessment | 30 days, 6 months,and 12 months
  SF-12
NYHA function | 7 days or discharge, 30 days, 6 months ,12 months and 2-5 years
Rate of All-cause Mortality | Immediate post- procedure ,7 days /discharge, 30 days, 6 months and 2-5 years.
Incidence of Myocardial Infarction | Immediate post- procedure, 7 days /discharge, 30 days, 6 months ,12months and 2-5 years.
Incidence of MACCE(including mortality, stroke, MI, re-procedure, Conduction disturbances and cardiac arrhythmias) | Immediate post- procedure, 7 days /discharge, 30 days, 6 months,12months and 2-5 years.
Incidence of Bleeding (life-threatening or disabling and major) | Immediate post- procedure, 7 days /discharge, 30 days, 6 months,12months and 2-5 years.
Incidence of Stroke | 7 days /discharge, 30 days, 6 months, 12 months and 2-5 years.
Incidence of AKI (stage 2 and 3,or renal replacement therapy (RRT: Hemodialysis, abdomen Cavity dialysis, hemofiltration)) | 7 days /discharge, 30 days, 6 months, 12 months and 2-5 years.
Incidence of Permanent Pacemaker Implantation | 7 days /discharge, 30 days, 6 months, 12 months and 2-5 years.
Incidence of major vascular complications | Immediate post- procedure, 7 days /discharge, 30 days, 6 months, 12 months.
Incidence of Conduction disturbances and cardiac arrhythmias | Immediate post- procedure, 7 days /discharge, 30 days, 6 months, 12 month and 2-5years
Incidence of Other TAVI-related Complications | Immediate post- procedure, 7 days /discharge, 30 days, 6 months, 12 month and 2-5years
  including transfer to surgery , Accidental heart-lung machine, coronary obstruction, ventricular septal rupture, Mitral valve damage or dysfunction，cardiac tamponade，endocarditis ，valvular thrombus，Valve migration(shifting, detachment,embolism,error deployment）,valve in valve

CONTACTS AND LOCATIONS:
Overall Officials: Yongjian Wu, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, CAMS&PUMC, Beijing, China

IPD SHARING:
Plan to Share IPD: No